CLINICAL TRIAL: NCT01870206
Title: Phase III Immunogenicity, Safety, Poliovirus Excretion and Acceptance of Vaccination OPV (Vero Cells) in Newborns Mexicans
Brief Title: Randomized Clinical Trial to Evaluate Immunogenicity and Safety in Mexicans Newborns
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios de Biologicos y Reactivos de México, S.A. de C.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: Birmex-ECA-01-2013
Record Dates: First submitted 2013-05-15; First posted 2013-06-05 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Poliomyelitis
Keywords: Immunogenicity; Safety; Efficacy; Poliomyelitis; Newborn
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trivalent OPV Birmex (Experimental): Newborns receive OPV vaccine produced in Vero cells by Birmex one dose of vaccine. A second dose four weeks after the first application.
  Interventions: Biological: Trivalent OPV Birmex
- Trivalent OPV Sanofi Pasteur (Active Comparator): Newborns who receive OPV vaccine produced in Vero cells by Sanofi Pasteur one dose of vaccine. A second dose four weeks after the first application.
  Interventions: Biological: Trivalent OPV Sanofi Pasteur

INTERVENTIONS:
Biological: Trivalent OPV Birmex — Newborns who receive OPV vaccine produced in Vero cells by Birmex one dose of vaccine immediately after random allocation (at birth). A second dose is given four weeks after the first application.
  Other Names: tOPV
  Arms: Trivalent OPV Birmex
Biological: Trivalent OPV Sanofi Pasteur — Newborns who receive OPV vaccine produced in Vero cells by Sanofi Pasteur one dose of vaccine immediately after random allocation (at birth). A second dose is given four weeks after the first application.
  Other Names: tOPV
  Arms: Trivalent OPV Sanofi Pasteur

SUMMARY:
Polio is a highly infectious disease caused by a virus. It invades the nervous system, and can cause total paralysis in a matter of hours. The virus enters the body through the mouth and multiplies in the intestine. Initial symptoms are fever, fatigue, headache, vomiting, stiffness in the neck and pain in the limbs. One in 200 infections leads to irreversible paralysis (usually in the legs). Among those paralysed, 5% to 10% die when their breathing muscles become immobilized. There is no cure for polio, it can only be prevented. Polio vaccine, given multiple times, can protect a child for life.

Compare in newborns the immunogenicity and safety of the vaccine OPV produced by Birmex compared with the vaccine OPV produced by Sanofi Pasteur, both produced in Vero cells.

DETAILED DESCRIPTION:
This is a randomized clinical trial, which includes 320 newborns of both sexes and residents of the state of México, 160 newborns receive the vaccine OPV Birmex and 160 newborns receive the vaccine OPV Sanofi Pasteur

ELIGIBILITY:
Inclusion Criteria:

* Newborns babies
* Weight ≥ 2.5 kg
* Have not received any doses of Polio Vaccine
* Whose parents or guardians reside in the work area
* Whose parent or guardian accept to sign written informed consent (by the other, father or guardian).

Exclusion Criteria:

* Born of a high-risk pregnancy.
* Weight ≤ 2.5 kg
* Presence of fever, diarrhea, known immunosuppression, respiratory infections.
* Treatment with immunosuppressants.
* Having neurological diseases.
* Require or received surgery in oropharynx.

Ages: 1 Day to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change seroconversion after one dose of trivalent vaccine OPV | after the first dose is taken blood samples (baseline, 30 and 60 days)

SECONDARY OUTCOMES:
Evaluate the adverse events in newborns babies | inmediately after treatment and during 60 days

OTHER OUTCOMES:
Poliovirus Excretion | Evaluate viral excretion rate, basal 7, 14, 21 and 28 days after vaccination of two vaccines against polio OPV in newborns Mexicans

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Rodríguez Álvarez, PhD, Principal Investigator — Laboratorios de Biológicos y Reactivos de México S.A de C.V
Locations (1):
- Hospital General de Chalco Dr. Fernando Quiroz Gutierrez, Valle de Chalco, State of Mexico, Mexico

REFERENCES:
- See also: Laboratorios de Biológicos y Reactivos de México S.A de C.V — http://www.birmex.gob.mx